CLINICAL TRIAL: NCT01568359
Title: Calcium Homeostasis in Acromegaly: Effect of Surgical/Medical Treatment and Comparison With Nonfunctioning Pituitary Tumors.
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Adriana Ioachimescu, MD, PhD, Associate Professor, Emory University
Other Study IDs: IRB00046786
Record Dates: First submitted 2012-03-29; First posted 2012-04-02 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Acromegaly; Nonfunctioning Pituitary Tumor
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine samples obtained from subjects.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1 - Acromegaly, Group 2 - control: Group 1 - Acromegaly patients, Group 2 - Nonfunctioning pituitary adenoma patients (control)

SUMMARY:
The purpose of the study is to evaluate the Calcium homeostasis in adult patients with uncontrolled acromegaly. The measurements will be repeated 3-6 months after the treatment of acromegaly (surgical or medical). The control group consists of patients with nonfunctioning pituitary tumors who will undergo surgical removal.

DETAILED DESCRIPTION:
Calcitriol is the active form of vitamin D. Parathyroid hormone (PTH) is secreted by the parathyroid glands in the neck. Both these chemicals are responsible for keeping the levels of calcium and phosphorous normal and also play a role in bone health. They can be measured in the blood. In some disorders, PTH or calcitriol levels are elevated, which results in increased calcium absorption from the gut, increased calcium in the bloodstream, and increased calcium excretion in the urine. Increased calcium in the urine can lead to the development of kidney stones. Increased calcium in the bloodstream can have adverse effects on the heart, gut, kidneys, and bones.

Acromegaly is a condition where a pituitary tumor secretes excessive amounts of growth hormone. Patients with acromegaly have been found to have a higher prevalence of kidney stones, urinary calcium, and serum calcium when compared to normal adults. The reason for this is unknown but a suggested mechanism is that growth hormone stimulates the production of calcitriol or PTH. If this is true, then treatment of acromegaly resulting in lower growth hormone levels should also result in lower blood and urine calcium levels. The investigators want to see if patients with acromegaly have high calcitriol, and vitamin D binding protein, or PTH levels and see if they change after treatment of the condition. The investigators also want to assess the amount of calcium in the urine, before and after treatment.

Patients with acromegaly may have disorders of bone health. The reason for this is unknown but a suggested mechanism is that growth hormone affects bone remodeling. The investigators want to see if patients with acromegaly have abnormal bone markers, specifically PINP, CTX, and TRAP, and to see if they change after treatment of the condition.

In order to see if the results are specific to patients with acromegaly, the investigators also want to check these levels in patients who do not have acromegaly, but have a "nonfunctioning" pituitary tumor. A nonfunctioning pituitary tumor is one that does not secrete excessive hormones in the bloodstream.

The specific aims of this study are:

1. To describe baseline calcitriol/PTH status in patients with uncontrolled acromegaly.
2. To assess the change in calcitriol/PTH levels after treatment with acromegaly (surgical or medical).
3. To evaluate the calcium and calcitriol/PTH levels in patients with acromegaly compared to patients with nonfunctioning pituitary adenomas.

This is a voluntary study. Adult patients with a diagnosis of acromegaly or a clinically nonfunctioning pituitary tumor receiving treatment at the Emory University Pituitary center will be given the opportunity to enroll in the study. Those that agree to participate will need to give written informed consent. Approximately 3 tablespoons (44ml) of blood will be drawn at enrollment for testing of vitamin D status and parathyroid hormone. If patients are already undergoing a blood draw for standard laboratory tests, then the volume of 44ml of blood will be obtained at the same time in order to avoid an additional needle stick. In addition, a 24-hour urine collection will be obtained to assess the amount of calcium present in the urine. Please note that medical or surgical therapy for your pituitary condition is determined by your endocrinologist and/or neurosurgeon and not part of the research study.

Within 6 months after treatment for pituitary treatment is initiated, when patients return to Emory University pituitary clinic for routine visit, laboratory data (vitamin D and parathyroid hormone) and repeat urine studies (24 hour urine collection) will be collected.

The confidentiality will be respected in all encounters. No personal identifiers are disclosed in any publications. Hard copy data will be kept securely in a locked office building with limited access and electronic data will always be password protected with access available to study personnel only. If abnormal results are discovered as part of testing done for this study, those results will be released to the patient's primary physician. All patients will be undergoing standard therapy for their pituitary disorder.

Results of this study may have important implications for future studies that are designed to evaluate the mechanism of how growth hormone may increase calcitriol levels.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with acromegaly or a nonfunctioning pituitary who will receive treatment for the pituitary condition.
* Study subjects must agree to participate in this study and provide written consent.
* Site- Emory Clinic/Emory University hospital.
* Stage of Disease: Patients with active acromegaly that is either newly diagnosed or uncontrolled on current therapy (as shown by GH/IGF-1 levels). Patients with nonfunctioning pituitary adenoma in whom surgical intervention planned based on current guidelines will serve as a control group.
* Age: Study subjects must be over 18 years of age.

Exclusion Criteria:

* Age < 18 years old
* Prior other diseases: Patients chronic renal disease stage 3 or worse (estimated GFR > 60).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with uncontrolled acromegaly and nonfunctioning pituitary adenomas presenting to the Emory University Pituitary Center for medical or surgical treatment.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2011-12; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Calcitriol/PTH | Baseline and 3-6 months after trreatment of pituitary condition
  To describe baseline calcitriol/PTH status in patients with uncontrolled acromegaly, with subanalyses based on presence of hyperprolactinemia.
  To assess the change in calcitriol/PTH levels after treatment with acromegaly, with subanalyses based on type of therapy (surgical or medical).
  To evaluate the calcium and calcitriol/PTH levels in patients with acromegaly compared to patients with nonfunctioning pituitary adenomas, with subanalyses based on presence of hyperprolactinemia in either group.

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Ioachimescu, MD, PhD, Principal Investigator — Asst Professor
Locations (2):
- United States (2):
  - Emory Clinic, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia

REFERENCES:
- [Background] Wongsurawat N, Armbrecht HJ, Zenser TV, Forte LR, Davis BB. Effects of hypophysectomy and growth hormone treatment on renal hydroxylation of 25-hydroxycholecalciferol in rats. J Endocrinol. 1984 Jun;101(3):333-8. doi: 10.1677/joe.0.1010333. PMID 6610018
- [Background] Ajibade DV, Dhawan P, Fechner AJ, Meyer MB, Pike JW, Christakos S. Evidence for a role of prolactin in calcium homeostasis: regulation of intestinal transient receptor potential vanilloid type 6, intestinal calcium absorption, and the 25-hydroxyvitamin D(3) 1alpha hydroxylase gene by prolactin. Endocrinology. 2010 Jul;151(7):2974-84. doi: 10.1210/en.2010-0033. Epub 2010 May 12. PMID 20463051
- [Background] Charoenphandhu N, Wongdee K, Krishnamra N. Is prolactin the cardinal calciotropic maternal hormone? Trends Endocrinol Metab. 2010 Jul;21(7):395-401. doi: 10.1016/j.tem.2010.02.002. Epub 2010 Mar 20. PMID 20304671
- [Background] Lancer SR, Bowser EN, Hargis GK. The effect of growth hormone on parathyroid function in rats. Endocrinology. 1976 May;98(5):1289-93. doi: 10.1210/endo-98-5-1289. PMID 1261522
- [Background] Cook DM, Ezzat S, Katznelson L, Kleinberg DL, Laws ER Jr, Nippoldt TB, Swearingen B, Vance ML; AACE Acromegaly Guidelines Task Force. AACE Medical Guidelines for Clinical Practice for the diagnosis and treatment of acromegaly. Endocr Pract. 2004 May-Jun;10(3):213-25. doi: 10.4158/EP.10.3.213. No abstract available. PMID 15382339
- [Background] Ezzat S, Melmed S, Endres D, Eyre DR, Singer FR. Biochemical assessment of bone formation and resorption in acromegaly. J Clin Endocrinol Metab. 1993 Jun;76(6):1452-7. doi: 10.1210/jcem.76.6.8501150.
- [Background] Nadarajah A, Hartog M, Redfern B, Thalassinos N, Wright AD, Joplin GF, Fraser TR. Calcium metabolism in acromegaly. Br Med J. 1968 Dec 28;4(5634):797-801. doi: 10.1136/bmj.4.5634.797. PMID 5702295
- [Background] Sigurdsson G, Nunziata V, Reiner M, Nadarajah A, Joplin GF. Calcium absorption and excretion in the gut in acromegaly. Clin Endocrinol (Oxf). 1973 Jul;2(3):187-92. doi: 10.1111/j.1365-2265.1973.tb00418.x. No abstract available. PMID 4760543
- [Background] Takamoto S, Tsuchiya H, Onishi T, Morimoto S, Imanaka S, Mori S, Seino Y, Uozumi T, Kumahara Y. Changes in calcium homeostasis in acromegaly treated by pituitary adenomectomy. J Clin Endocrinol Metab. 1985 Jul;61(1):7-11. doi: 10.1210/jcem-61-1-7. PMID 3839000
- [Background] Halse J, Haugen HN. Calcium and phosphate metabolism in acromegaly. Acta Endocrinol (Copenh). 1980 Aug;94(4):459-67. doi: 10.1530/acta.0.0940459. PMID 6254298
- [Background] Hennessey JV, Jackson IM. Clinical features and differential diagnosis of pituitary tumours with emphasis on acromegaly. Baillieres Clin Endocrinol Metab. 1995 Apr;9(2):271-314. doi: 10.1016/s0950-351x(95)80338-6. PMID 7625986
- [Background] Brown DJ, Spanos E, MacIntyre I. Role of pituitary hormones in regulating renal vitamin D metabolism in man. Br Med J. 1980 Feb 2;280(6210):277-8. doi: 10.1136/bmj.280.6210.277. PMID 7357340
- [Background] White HD, Ahmad AM, Durham BH, Chandran S, Patwala A, Fraser WD, Vora JP. Effect of active acromegaly and its treatment on parathyroid circadian rhythmicity and parathyroid target-organ sensitivity. J Clin Endocrinol Metab. 2006 Mar;91(3):913-9. doi: 10.1210/jc.2005-1602. Epub 2005 Dec 13. PMID 16352693
- [Background] Lund B, Eskildsen PC, Lund B, Norman AW, Sorensen OH. Calcium and vitamin D metabolism in acromegaly. Acta Endocrinol (Copenh). 1981 Apr;96(4):444-50. doi: 10.1530/acta.0.0960444. PMID 7211102
- [Background] Parkinson C, Kassem M, Heickendorff L, Flyvbjerg A, Trainer PJ. Pegvisomant-induced serum insulin-like growth factor-I normalization in patients with acromegaly returns elevated markers of bone turnover to normal. J Clin Endocrinol Metab. 2003 Dec;88(12):5650-5. doi: 10.1210/jc.2003-030772. PMID 14671148
- [Background] Chanson P, Salenave S, Kamenicky P, Cazabat L, Young J. Pituitary tumours: acromegaly. Best Pract Res Clin Endocrinol Metab. 2009 Oct;23(5):555-74. doi: 10.1016/j.beem.2009.05.010. PMID 19945023
- [Derived] Constantin T, Tangpricha V, Shah R, Oyesiku NM, Ioachimescu OC, Ritchie J, Ioachimescu AG. Calcium and Bone Turnover Markers in Acromegaly: A Prospective, Controlled Study. J Clin Endocrinol Metab. 2017 Jul 1;102(7):2416-2424. doi: 10.1210/jc.2016-3693. PMID 28407138